CLINICAL TRIAL: NCT06546358
Title: A Pilot, Double-blind, Randomized Trial of Quetiapine Versus Trazadone in Women With Postpartum Depression
Brief Title: Quetiapine Versus Trazadone in Women With Postpartum Depression
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 125638
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; trazadone; quetiapine
MeSH Terms: conditions — Depression, Postpartum | interventions — Trazodone; Quetiapine Fumarate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to treatment with trazodone or quetiapine in blocks of 8 with a sequence generated by SPSS.
Who Masked: Participant
Masking Description: Pharmacy will randomize and dispense medication. Participants will be started on trazodone 12.5 mg or quetiapine 6.25 mg in identical opaque gelatin capsules at bedtime.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trazadone (Active Comparator): Participants will be started on trazodone 12.5 mg or quetiapine 6.25 mg in identical opaque gelatin capsules at bedtime. The doses will be increased to a maximum of 50 mg for trazodone and 25 mg for quetiapine.
  Interventions: Drug: Trazodone
- Quetiapine (Active Comparator): Participants will be started on trazodone 12.5 mg or quetiapine 6.25 mg in identical opaque gelatin capsules at bedtime. The doses will be increased to a maximum of 50 mg for trazodone and 25 mg for quetiapine.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Trazodone — Participants will be randomized to receive either quetiapine or trazodone.
  Other Names: Teva-Trazadone
  Arms: Trazadone
Drug: Quetiapine — Participants will be randomized to receive either quetiapine or trazodone.
  Other Names: Quetiapine Fumarate
  Arms: Quetiapine

SUMMARY:
Postpartum depression is a serious disorder that affects approximately 17% of women who have recently given birth. Untreated postpartum depression can negatively affect the mother, the infant, and the family. Lack of sleep is common after delivery and can trigger or worsen depression in some women. Trazodone is used for sleeplessness and depression, but it has not been studied for postpartum depression. There is preliminary evidence that quetiapine, another drug used for depression and sleeplessness, may be effective for postpartum depression. We are planning a study to compare the effectiveness and side effects of quetiapine and trazodone in women with postpartum depression. The results of this study will help us carry out larger studies comparing these drugs with a placebo (a sugar pill) in postpartum depression. We expect the results of our study will improve the mental health of mothers and the well-being of their babies and make it easier for healthcare staff to select the right drug for women with postpartum depression.

DETAILED DESCRIPTION:
Design: This double-blind, flexible dosing study aims to compare the effectiveness and tolerability of trazodone and quetiapine in women with PPD. The study will be conducted at the Parkwood Institute Mental Health Care after obtaining approval from the Western University Health Sciences Research Ethics Board. Since trazodone and quetiapine are not indicated for the treatment of PPD, approval will also be obtained from Health Canada. Patients will receive written and verbal information about the study and informed consent will be obtained before study participation. Participants: Outpatients between ages 18 and 45 years who are within 6 months of delivering a child and have a DSM-5-TR diagnosis of major depressive disorder (MDD) with peripartum onset, a 17-item Hamilton Depression Rating Scale (HDRS) score of >18 at both the screening and baseline visits, can communicate in English, and can provide informed consent will be included. Because women remain at risk for the occurrence of depression for several weeks after delivery, the peripartum onset will be changed to 3 months after delivery rather than the DSM-5-TR recommended 4 weeks duration. Exclusion criteria: Women with schizophrenia spectrum or other psychotic disorders, bipolar and related disorders, eating disorders, substance-related and addictive disorders; and those at high risk for suicide (actively suicidal or with a score of ≥ 3 on item #3 on the HDRS) will be excluded. Women with a physical illness that is a contraindication to the use of quetiapine, or who have a history of intolerance or nonresponse to quetiapine will also be excluded. Assessment and schedule: The schedule of assessments for each participant is outlined in Appendix I. Participants will be randomized in a 1:1 ratio to treatment with trazodone or quetiapine in blocks of 8 with a sequence generated by SPSS. Participants will be started on trazodone 12.5 mg or quetiapine 6.25 mg in identical opaque gelatin capsules at bedtime. The doses will be increased to a maximum of 50 mg for trazodone and 25 mg for quetiapine. Follow-up visits will be scheduled for weeks 1, 2, 4, 6, and 8 weeks.

The primary outcome will be the mean change from baseline to week 8 in the HDRS total score, the proportion of participants achieving response (≥50% reduction in HDRS score at baseline), and the proportion of participants achieving remission (HDRS ≤12). The mean change in scores of the Edinburgh Postnatal Depression Scale (EPDS), Generalized Anxiety Disorder 7-item (GAD-7) scale, Young Mania Rating Scale (YMRS), and the Barkin Index of Maternal Functioning (BIMF) from baseline to week 8 will also be assessed. Safety measures include measurement of blood pressure, pulse rate, body weight, CBC, ECG, TSH, and pregnancy test. The Frequency, Intensity, Burden of Side Effects Rating scale (FIBSER) will be used to gather information about the side effects of trazodone and quetiapine. The BIMF will assess maternal functioning. Since the postpartum period is also associated with the first onset of hypo/mania, participants will be assessed using the YMRS. Following study completion or discontinuation from the study, any serious adverse events or side effects that caused study discontinuation will be followed up. Adherence will be determined by the returned tablet count.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between ages 18 and 45 years who are within 6 months of delivering a child and have a DSM-5-TR diagnosis of major depressive disorder (MDD) with peripartum onset, a 17-item Hamilton Depression Rating Scale (HDRS) score of >18 at both the screening and baseline visits, can communicate in English, and can provide informed consent will be included.

Exclusion Criteria:

* Women with schizophrenia spectrum or other psychotic disorders, bipolar and related disorders, eating disorders, substance-related and addictive disorders; and those at high risk for suicide (actively suicidal or with a score of ≥ 3 on item #3 on the HDRS) will be excluded. Women with a physical illness that is a contraindication to the use of quetiapine, or who have a history of intolerance or nonresponse to quetiapine will also be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women will be recruited who have given birth within the last 6 months.
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 8 weeks
  The primary outcome will be the mean change from baseline to week 8 in the HDRS total score, the proportion of participants achieving response (≥50% reduction in HDRS score at baseline), and the proportion of participants achieving remission (HDRS ≤12).

CONTACTS AND LOCATIONS:
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data is available upon request.